CLINICAL TRIAL: NCT06975410
Title: A Phase 1/2, Open-label, Multicenter, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of YH32364 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Clinical Trial of YH32364 in Patients With Locally Advanced or Metastatic EGFR Overexpressing Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH32364-101
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: EGFR Overexpression; Locally Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: YH32364; EGFR/4-1BB bispecific antibody; Solid tumor; Head and neck squamous cell carcinoma (HNSCC); Non-small cell lung cancer (NSCLC); Esophageal squamous cell carcinoma (ESCC); Biliary tract cancer (BTC); Uterine cervical cancer; Vulvar cancer; Urothelial cancer
MeSH Terms: conditions — Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Esophageal Squamous Cell Carcinoma; Biliary Tract Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YH32364 (Experimental): Dose Escalation Part: Dose Escalation part is designed to assess the safety and tolerability of YH32364 and to identify the Maximum Tolerated dose (MTD) and/or two dose levels for recommended dose (RD) selection.
  Dose Expansion Part: Dose Expansion part will consist of multiple cohorts by cancer types. Cohort 1 will be initiated to determine the RD after completion of Part 1. The RD will be determined among two dose levels investigated in Cohort 1 based on the totality of available data including PK, biomarkers, dose-response, safety, and efficacy.
  Interventions: Drug: YH32364

INTERVENTIONS:
Drug: YH32364 — Dose Escalation Part: In this part, 6 dose levels are planned and approximately 30 patients will be enrolled. After each dose level, Safety Review Committee (SRC) will evaluate the available safety, tolerability, PK of YH32364 to decide the next dose.
  Dose Expansion Part: 50 participants with previously treated locally advanced or metastatic EGFR overexpressing HNSCC other than NPC will be randomized 1:1 ratio to each dose. (Cohort 1: Participants with locally advanced or metastatic EGFR overexpressing HNSCC other than NPC, whose disease progressed after or who are intolerable to all the available standard treatment)

SUMMARY:
This is a study for people with locally advanced or metastatic cancer for whom previous treatment was not successful. Adults aged 18 and over with advanced cancer with Epidermal Growth Factor Receptor (EGFR) overexpressing can join the study. The purpose of this study is to find out whether a medicine called YH32364 helps people with locally advanced or metastatic cancers with EGFR overexpression.

DETAILED DESCRIPTION:
YH32364 is a new type of immunotherapy called a bispecific antibody that targets both Epidermal Growth Factor Receptor (EGFR) and 4-1BB. EGFR is a gene involved in cancer growth, and many cancer treatments aim to target it. 4-1BB, an immune-modulating protein, plays an important role in boosting T cell activity to combat cancer.

YH32364 is a treatment designed to activate 4-1BB specifically in tumors, aiming to avoid the liver-related side effects seen with previous 4-1BB treatments. It also helps block EGFR signals, assumed to make EGFR-targeted therapies more effective by overcoming resistance.

This study is consists of two parts. In Part 1, participants will be assigned sequentially to one of six dose levels, ranging from the lowest to the highest dose as determined by the sponsor, in order to identify an appropriate dosage.

In Part 2, participants will be randomly assigned to one of the two optimal dose levels identified in Part 1 to confirm the recommended dose.

The YH32364 will be administered via intravenous (IV) infusion once every two weeks. Participants will be required to visit the study site regularly for treatment and assessments. During all the visits, the doctors check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form (ICF) prior to any study specific procedures
* ECOG performance status 0 or 1
* Estimated life expectancy of at least 3 months
* A woman must not be breastfeeding
* Have at least one measurable lesion, not previously irradiated and not chosen for biopsy during the study screening period, that can be accurately measured at baseline ≥10 mm in the longest diameter (except lymph nodes which must have a short axis of ≥15 mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), are suitable for accurate repeated measurements.

[Dose Escalation Only] Locally advanced or metastatic EGFR overexpressing solid tumor* that is refractory or intolerable on all available standard therapy and that is considered uncurable by local therapy

* One of the following pathologically confirmed EGFR overexpressing (IHC3+ or IHC2+) tumors.

* Head and neck squamous cell carcinoma (HNSCC)
* Non-small cell lung cancer (NSCLC): squamous cell carcinoma (SqCC)
* Esophageal squamous cell carcinoma (ESCC)
* Biliary tract cancer (BTC)
* Uterine cervical cancer
* Vulvar cancer
* Urothelial cancer
* Squamous cell carcinoma of other origin of tumor (e.g., skin squamous cell tumor)

[Dose Expansion Only] Cohort 1: Pathologically confirmed EGFR overexpressing (IHC3+ or IHC2+), locally advanced or metastatic HNSCC other than nasopharyngeal carcinoma (NPC)* that is refractory or intolerable on all available standard therapy and that is considered uncurable by local therapy.

Exclusion Criteria:

* Known uncontrolled central nervous system (CNS) metastases, spinal cord compression, and/or carcinomatous meningitis
* Have history of a second primary cancer with the exception of

  * curatively treated non-melanomatous skin cancer
  * curatively treated cervical or breast carcinoma in situ, or
  * other malignancy with no known active disease present and no treatment administered during the last 2 years
* Have history of or current Class II, III or IV heart failure as defined by the New York Heart Association (NYHA)
* Have history of acute coronary syndromes, including myocardial infarction, coronary artery bypass graft, unstable angina, coronary angioplasty or stenting within past 24 weeks
* Have history of (non-infectious) interstitial lung disease (ILD) or pneumonitis that required steroids, or any evidence of current ILD or pneumonitis
* Have autoimmune disease that has required systemic treatment
* Infection with human immunodeficiency virus (HIV)
* Active chronic hepatitis B or chronic hepatitis C

[Prior/Concomitant Therapy]

* Have received systemic steroid therapy
* Previous treatment with a 4-1BB/CD137-modulating agent
* Have used a live vaccine within 4 weeks
* Have received treatment with immunotherapy, biological therapies, targeted small molecules, or hormonal therapies
* Have received radiation therapy
* Have received cytotoxic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) including dose limiting toxicities (DLTs) | Study Day 1 to Study Day 28 (during the DLTs evaluation period)
  To assess the safety and tolerability of YH32364 in order to determine maximum tolerated dose (MTD) and select doses for dose optimization
Objective Response Rate (ORR) | through dose expansion part completion, approximately 1.5 year
  To assess the ORR of YH32364 at the recommended dose (RD) according to RECIST v1.1 by Investigator assessment

SECONDARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
AUC from time 0 to infinity (AUCinf) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Maximum observed serum concentration (Cmax) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Time to reach Cmax (Tmax) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Apparent terminal elimination half-life (t1/2) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Total clearance (CL) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Volume of distribution (Vd) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Volume of distribution at steady state (Vss) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
AUC during dosing interval at steady state (AUCtau) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Cmax at steady state (Cmax,ss) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Time to reach Cmax,ss (Tmax,ss) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Accumulation ratio (Rac) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Trough (predose) serum concentration on Cycle 4 (Ctrough) | through study completion, approximately 2.5 year
  To characterize the pharmacokinetics (PK) of YH32364
Presence and characterization of YH32364 ADA including neutralizing antibodies | through study completion, approximately 2.5 year
  To explore the immunogenicity of YH32364
Titer of YH32364 ADA | through study completion, approximately 2.5 year
  To explore the immunogenicity of YH32364
Objective Response Rate (ORR) | through dose escalation part completion, approximately 1 year
  To assess the anti-tumor activity according to RECIST v1.1 by Investigator assessment
Duration of Response (DoR) | through study completion, approximately 2.5 year
  To assess the anti-tumor activity according to RECIST v1.1 by Investigator assessment
Disease Control Rate (DCR) | through study completion, approximately 2.5 year
  To assess the anti-tumor activity according to RECIST v1.1 by Investigator assessment
Depth of Response | through study completion, approximately 2.5 year
  To assess the anti-tumor activity according to RECIST v1.1 by Investigator assessment
Time to Response | through study completion, approximately 2.5 year
  To assess the anti-tumor activity according to RECIST v1.1 by Investigator assessment
Progression-free survival (PFS) | through study completion, approximately 2.5 year
  To assess the anti-tumor activity according to RECIST v1.1 by Investigator assessment
TEAEs | through dose expansion part completion, approximately 1.5 year
  To assess the safety and tolerability of YH32364
Overall Survival (OS) | through dose expansion part completion, approximately 1.5 year
  To assess the overall survival of YH32364 at the RD

OTHER OUTCOMES:
Immune ORR (iORR) | through study completion, approximately 2.5 year
  To assess the immune-related efficacy according to iRECIST by Investigator assessment
Immune Duration of Response (iDOR) | through study completion, approximately 2.5 year
  To assess the immune-related efficacy according to iRECIST by Investigator assessment
Immune PFS (iPFS) | through study completion, approximately 2.5 year
  To assess the immune-related efficacy according to iRECIST by Investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Yuhan Clinical Research Physician, Study Director — Yuhan Corporation
Locations (4):
- South Korea (4):
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to clinicaltrials@yuhan.co.kr
  A summary of the study results will be posted in the publicly accessible database (i.e. clinicaltrials.gov) no later than 1 year after the study's primary completion date.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 1 year and ending 5 years after all trial endpoints were assessed
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to clinicaltrials@yuhan.co.kr